CLINICAL TRIAL: NCT02928913
Title: The Associations Between Sedentary Behaviour and Impact Characteristics on Bone Health
Status: Completed | Type: Observational
Sponsor: Dr Tina Smith (Other)
Collaborators: London South Bank University (Other)
Responsible Party: Sponsor-Investigator, Dr Tina Smith, Senior Lecturer in Biomechanics, University of Wolverhampton
Organization: University of Wolverhampton (Other)
Other Study IDs: 01/0416/TS/UOW
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Bone Health
Keywords: sedentary; non-sedentary; populations
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sedentary: Predominantly engage in sedentary behaviours
  Interventions: Other: No intervention
- Non-sedentary: Predominantly engage in non-sedentary behaviours
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
To investigate associations between sedentary and active behaviour with bone health and functional ability, and to associate mechanical loading at the lumbar spine and hip in sedentary and active individuals with bone mineral density.

DETAILED DESCRIPTION:
Significant proportions of adults engage in sedentary behaviour for prolonged periods of time which is generally regarded as having deleterious effects on health. However, far less is known about its specific effects on bone health. Exercise has been proposed as a method of improving bone health, as impact forces generated as the foot contacts the ground during physical activity have the potential to aid bone maintenance and development.

The properties of bone are regulated through the amount mechanical loading, frequency of loading and duration of loading endured, which can create an osteogenic effect. These variables can be quantified via accelerometry which records the magnitude, rate and duration of accelerations experienced at the site on the body where the accelerometer is worn. Although there is a vast amount of literature where accelerometers have been used to monitor physical activity, there is a lack of studies that use accelerometers to determine the most effective exercise for bone, especially in relation to the lumbar spine. Exploring the bone health and loading characteristics of sedentary and low and highly active non-sedentary individuals will provide evidence upon which to base future interventions that are likely to be of benefit for bone health in sedentary populations.

ELIGIBILITY:
Inclusion Criteria:

Male or female aged 30 - 60 years Individuals who are sedentary and do not participate in physical activities Individuals who participate in some physical activities Individuals who are highly active Must be free from injury or illness that will affects following typical weekly routines.

Exclusion Criteria:

Any medical condition that affects bone health, e.g. osteoporosis. Currently takes medication that affects bone health, e.g. long term steroid use.

Inability to participate in typical daily activity, e.g. severe arthritis, injury. Women who are post menopause Women who are on hormone replacement therapy Unable to participate in DXA scan, e.g. due to recent exposure to radiation, pregnancy status.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sedentary and non-sedentary populations.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | One day

SECONDARY OUTCOMES:
Mechanical loading dose during daily activity via accelerometry | 7 days
Mechanical loading intensity during daily activity via accelerometry | 7 days
Functional movement assessment: Grip Strength | One day
Functional movement assessment: Timed up and go | One day
Functional movement assessment: 10m walk test | One day
Functional movement assessment: 5 times sit to stand | One day
Functional movement assessment: gait analysis (acceleration at hip and lumbar spine) | One day
Functional movement assessment: gait analysis (ground reaction force) | One day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wolverhampton, Walsall, West Midlands, United Kingdom